CLINICAL TRIAL: NCT00308659
Title: Diagnostic Strategy Evaluation Study of Two Diagnostic Strategies for the Treatment of SCAP : Noninvasive Strategy and Semiinvasive Strategy Including FOB Distal Samplings
Brief Title: Study to Evaluate Two Diagnostic Strategies for the Treatment of Severe Community Acquired Pneumonia (SCAP)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: SCAP FOB; CNMR grant, cardiff
Record Dates: First submitted 2006-03-28; First posted 2006-03-30 (Estimated); Last update posted 2006-03-30 (Estimated); Status verified 2006-03

CONDITIONS: Community Aquired Pneumonia

INTERVENTIONS:
Procedure: FOB protected distal microbiological samplings

SUMMARY:
Main hypothesis: microbiological diagnossis off severe community acquired pneumonia can be performed by non invasive or semi invasive microbiological tools, semi invasive tools including protected distal bronchial samplings by the mean of Fiber optic bronchoscopy (FOB). A microbiological diagnosis could improve antibiotic therapy efficacy and improve patient's outcome.

These Two strategies have never been prospectivally evauated.

* Aim of the study: To evaluate 2 diagnostic strategies: non invasive or semi invasive including protected distal bronchial samplings by the mean of Fiber optic bronchoscopy (FOB)for the care of patients admitted in intensive care for severe community acquired pneumonia and receiving an empirical antibiotic therapy as recommanded by 2001 American thoracic guidelines
* Type of study randomized multicentric controlled open study

DETAILED DESCRIPTION:
Type of study randomized multicentric controlled open study

Number of patients: 200 patients (100 patients in each group)admitted in ICU for SCAP

* Number of center : 5
* Clinical strategies under evaluation :
* Group A: semi-invasive strategy: FOB within 24 hours after ICU admission
* Group B: non-invasive strategy: no FOB within 24 hours after ICU admission
* Evaluation criteria:

Main criteria: Changes in initial empirical antibiotic treatment according to microbiological results obtained in each group.

others

* FOB related complications
* Microbiological results
* Type of antibiotic treatment modifications
* ICU outcome and outcome at day 28
* Duration of antibiotic therapy and nimber of days without antibiotics at day 28 after inclusion

ELIGIBILITY:
Inclusion Criteria:

New radiological infiltrate SCAP clinical diagnosis admitted in ICU Admitted in hospital for less than 24 hours Aged 18 or older Signed informed consent

Exclusion Criteria:

Pregnancy Muribond patients Previuos hospitalisation within One month Neutropenia None HIV status

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2006-03

CONTACTS AND LOCATIONS:
Overall Officials: RABBAT Antoine, MD, Principal Investigator — APHP
Locations (1):
- Hotel dieu, Paris, France